

# Effet des échanges transfusionnels sur l'efficience cognitive des patients atteints de drépanocytose

## PROTOCOLE DE RECHERCHE NON INTERVENTIONNELLE IMPLIQUANT LA PERSONNE HUMAINE

Réf. promoteur: D24-P021 - IDRCB: 2024-A02851-46

Investigateur Principal Mr Hugo BISMUTH

Service de Neurologie

Hôpital : GHU Paris Psychiatrie & Neurosciences, site Sainte Anne

Tél: 0145658644

Courriel: <u>H.BISMUTH@ghu-paris.fr</u>

Responsables scientifiques Dr Pauline NARME

Psychologue-Neuropsychologue Professeur des Universités Université Paris Cité Tél: 0608983804

Courriel: pauline.narme@u-paris.fr

Pr David CALVET

Chef de Service de Neurologie et Unité

Neurovasculaire

GHU Paris Psychiatrie et Neurosciences -

Hôpital Sainte-Anne Tél : 0145658634

Courriel: d.calvet@ghu-paris.fr

Promoteur Groupe Hospitalier Universitaire Paris –

Psychiatrie & Neurosciences (GHU Paris),

Hôpital Sainte Anne

Représenté par Mr CHAPELLE Directeur de la recherche, de l'innovation, des

partenariats et de la coopération internationale

1, rue Cabanis – 75014 Paris

Structure chargée

du suivi de la recherche DRCI (Délégation à la Recherche Clinique et à

l'Innovation)

Docteur Khaoussou SYLLA,

Coordinateur Médical

La recherche a reçu un avis favorable du CPP XXXX en date du

#### Page de signature

## Protocole de recherche non-interventionnelle impliquant la personne humaine

Titre: Effet des échanges transfusionnels sur l'efficience cognitive des patients atteints de drépanocytose

Acronyme: DREPA-COG

Version n° du : V1.1 du 28/07/2025

Réf. Promoteur : D24-P021 IDRCB : 2024-A02851-46

## Investigateur Principal /Coordonnateur

## Mr Hugo BISMUTH

Psychologue-Neuropsychologue

Service de Neurologie Date : <u>H.BISMUTH@ghu-paris.fr</u> Signature :

**GHU** Paris

## Responsables scientifiques

#### **Dr Pauline NARME**

Psychologue-Neuropsychologue

Professeur des Universités Date : Université Paris Cité Signature :

Tél: 0608983804

Courriel: <a href="mailto:pauline.narme@u-paris.fr">pauline.narme@u-paris.fr</a>

#### Pr David CALVET

Chef de Service de Neurologie et Unité Date : Neurovasculaire Signature :

GHU Paris Psychiatrie et Neurosciences –

Hôpital Sainte-Anne Tél : 0145658634

Courriel: <u>d.calvet@ghu-paris.fr</u>

#### **Promoteur**

GHU Paris Psychiatrie & Neurosciences

Son Représentant : DRCI

**Dr Khaoussou SYLLA**Coordonnateur Médical

Date :
Signature :

Tél: 01 45 65 76 78

Courriel: K.SYLLA@ghu-paris.fr

## TABLE DES MATIÈRES

## **RESUME**

| 1. | JUSTIFICATION SCIENTIFIQUE DE LA RECHERCHE | 12 |
|---|---|---|
| 1.1.<br>1.2.<br>1.3.<br>1.4. | ÉTAT ACTUEL DES CONNAISSANCES RELATIVES AU DOMAINE CONCERNE | 14<br>14 |
| 2. | OBJECTIFS | 14 |
| 2.1.<br>2.2. | OBJECTIF PRINCIPALOBJECTIFS SECONDAIRES | |
| 3. | METHODE ET POPULATION | 15 |
| 3.1.<br>3.2.<br>3.3. | CRITERES D'EVALUATION DEROULEMENT DE LA RECHERCHE DUREE DE LA RECHERCHE : | 16 |
| 4. | RISQUES ET VIGILANCES | 18 |
| 5. | ASPECTS STATISTIQUES | 18 |
| 5.1.<br>5.2.<br>5.3. | Justification statistique de la taille de l'echantillon | 19 |
| 6. | GESTION DES DONNEES | 21 |
| 6.1.<br>6.2.<br>6.3<br>6.4 | Modalites de recueil des donnees | 21<br>21 |
| 7. | CONTROL DE LA QUALITE | 23 |
| 7.1<br>7.2<br>7.3<br>7.4<br>7.5 | Qualification des intervenants Qualite des données Archivage Gestion des non conformites Audit | 23<br>23 |
| 8. | ASPECTS ETHIQUES ET LEGAUX | 24 |
| 8.1<br>8.2<br>8.3<br>8.4<br>8.5<br>8.6<br>8.7<br>8.8<br>8.9 | ROLE DU PROMOTEUR. ENGAGEMENT DE RESPONSABILITES DE L'INVESTIGATEUR PRINCIPAL. MODALITES D'INFORMATION DES SUJETS. DEMANDE D'AVIS AU COMITE DE PROTECTION DES PERSONNES (CPP). INFORMATION DE L'AGENCE NATIONALE DE SECURITE DU MEDICAMENT (ANSM). TRAITEMENT DES DONNEES A CARACTERE PERSONNEL. RESPONSABILITES DE L'INVESTIGATEUR VIS-A-VIS DU PROMOTEUR. RAPPORT FINAL DE LA RECHERCHE. PROPRIETE DES DONNEES. | |
| 9. | REGLES RELATIVES A LA PUBLICATION | |
| 7.<br>10. | FINANCEMENT ET ASSURANCE | |
| | URCE DE FINANCEMENT | 26 |
| 11. | BIBLIOGRAPHIE | 26 |

## **RESUME**

| GENERALITES | |
|---|---|
| Date – N° version protocole | V1.0 du<br>26/05/2025 |
| Date – N° version note d'information | V1.0 du<br>26/05/2025 |
| Date – N° version questionnaires/trame des entretiens | V.1 du<br>19/05/2025 |

| Conformité de cette demande d'avis avec la procédure prévue II de l'<br>du CSP - Une réponse négative à l'un de ces 4 items signifie que vous r<br>cette procédure. | |
|---|---|
| Cette recherche comporte uniquement des données recueillies par questionnaire(s) ou entretien(s) : | Oui Non |
| Cette recherche n'a aucune conséquence pour les personnes participantes que ce soit en termes de sécurité ou de modification de la prise en charge habituelle : | Oui Non |
| Cette recherche est dénuée de risques et les inconvénients pour les personnes participantes à la recherche sont négligeables : | Oui Non |
| Le recueil et le traitement des données mis en œuvre dans cette recherche sont conformes à la méthodologie de la référence MR-003 homologuée par la CNIL : | Oui Non |

| Titre de la recherche | Effet des échanges transfusionnels sur l'efficience cognitive des patients atteints de drépanocytose |
|---|---|
| Acronyme | DREPA-COG |
| N° IDRCB | 2024-A02851-46 |

## **LISTE DES ABREVIATIONS**

VT : Vitesse de Traitement ET : Échanges Transfusionnels

AVC: Accident Vasculaire Cérébral

EVQ : Échelle de douleur FSS: Fatigue Severity Scale

HADS: Hospital Anxiety and Depression Scale

SDMT: Symbol Digit Modality Test

T-MoCA: Téléphone Montréal Cognitive Assesment

| I – INFOR | MATIONS ADMINISTRATRIVES |
|---|---|
| Promoteur | Groupe Hospitalier Universitaire Paris – Psychiatrie<br>& Neurosciences |
| Représenté par | Délégation à la Recherche Clinique et à l'Innovation (DRCI) Direction de la Recherche, de l'innovation, des Partenariats et de la Coopération internationale. Mr Marin CHAPELLE 1, rue Cabanis 75014 PARIS k.sylla@ghu-paris.fr |
| Thèses et travaux Universitaire<br>Responsable Scientifique | Professeur David CALVET Neurologue Service de neurologie D.CALVET@ghu-paris.fr GHU PARIS Docteur Pauline NARME Psychologue-Neuropsychologue Professeur des Universités pauline.narme@u-paris.fr Université Paris Cité 0608983804 |
| Investigateur Principal | Hugo BISMUTH Psychologue-Neuropsychologue Service de Neurologie H.BISMUTH@ghu-paris.fr GHU Paris |
| Nombre de centres | 6 |

## II - CONTEXTE ET JUSTIFICATION DE LA RECHERCHE : RATIONNEL PRESENTANT LE CONTEXTE ET LES HYPOTHESES DE LA RECHERCHE

La drépanocytose est la maladie génétique la plus répandue en France et dans le monde. C'est une maladie des globules rouges, plus particulièrement de l'hémoglobine, à l'origine d'une anomalie du transport de l'oxygène vers les différents organes.

L'amélioration de la prise en charge des complications aigues de la maladie a révélé l'existence de complications chroniques, en particulier neurologiques, qui sont responsables de la plus grande partie du handicap chez l'adulte.

Aux séquelles visibles des Accidents Vasculaires Cérébraux (AVC) s'ajoutent les troubles cognitifs, à l'origine de difficultés importantes chez les patients drépanocytaires. Les fonctions exécutives qui permettent la planification de nos actions et qui régulent notre comportement sont principalement atteintes ou touchées chez l'adulte drépanocytaire. La vitesse de traitement (VT) des informations semble particulièrement touchée.

Un des traitements de la maladie consiste à réaliser des saignées-transfusions (remplacer le sang malade par du sang sain à intervalles réguliers). Ce traitement a un intérêt majeur sur l'évolution de la maladie. Des données préliminaires suggèrent que les échanges transfusionnels (ET) pourraient avoir un effet bénéfique sur la cognition. L'objectif de notre étude vise à évaluer la vitesse de traitement des informations à différentes périodes du cycle d'échanges transfusionnels. Si le lien était confirmé, nous aurions ainsi un marqueur neurologique de la maladie simple à évaluer et reproductible tant pour la prise en charge clinique que pour le suivi dans les essais thérapeutiques.

| III - OBJE | CTIFS ET CRITERES DE JUGEMENT |
|---|---|
| A - Objectif principal de la<br>recherche et critère de<br>jugement principal | Objectif principal: évaluer l'effet des échanges transfusionnels sur la vitesse de traitement des informations des patients drépanocytaires Critère de jugement principal: la vitesse de traitement des informations comme marqueur de l'atteinte cérébrale de la drépanocytose. Test utilisé: SDMT (Symbol Digit Modality Test) version orale. |
| B - Objectif(s) secondaire(s)<br>de la recherche et critère(s)<br>de jugement secondaire(s)<br>éventuel(s) | Evaluer l'effet des échanges transfusionnels sur les différentes fonctions cognitives Identifier les facteurs prédictifs associés à la vitesse de traitement en fonction du cycle |

| IV – ORGANISATION DE L'ETUDE | |
|---|---|
| | Étude non interventionnelle sur une cohorte de patients atteints de drépanocytose en programme d'échange transfusionnel |
| | de diepariocytose en programme à centange mansiosionnei |
| <b>A</b> - Description<br>synthétique du<br>schéma<br>d'étude | Le patient est informé dans l'un des centres participant à l'étude et ne s'oppose pas à y participer. La passation de tests cognitifs se fait à trois temps distincts (T0/T1/T2). Il s'agit d'une évaluation neuropsychologique courte (20-25 minutes) réalisée en distanciel, par le biais de la visioconférence. T0: dans les 48h précédant l'échange transfusionnel; T1: 7 à 9 jours après l'échange transfusionnel; T2: dans les 48h précédant l'échange suivant. La batterie est composée des tests suivants: Symbol Digit Modality Test (SDMT, Smith, 1973), MoCA (version T-MoCA, Narsredin et al., 2005), subtest Mémoire des Chiffres de la WAIS-IV (Wechsler, 2008), Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983), Fatigue Severity Scale (FSS, Krupp et al., 1989, échelle de douleur (gradient de 1 à 10). |
| | Cette évaluation est réalisée de façon centralisée en visioconférence par un neuropsychologue formé à la passation de ces tests spécifiques. |
| <b>B</b> - Méthodologi<br>1 - Questionnaire<br>Modalités de po | |
| Questionnaire<br>administré par | Courrier Internet Téléphone |
| - Garriir iisire pai | Si autre préciser : visioconférence par le biais d'un ordinateur |
| Questionnaire<br>administré en | Une fois Plusieurs fois |
| dariiriisire eri | Si plusieurs fois préciser le nombre de passation : 3 |
| Type de<br>questionnaire | Validé Si validé indiquer le type de validation: les tests neuropsychologiques utilisés dans le protocole sont validés car ils ont fait l'objet de plusieurs études scientifiques démontrant leurs qualités psychométriques (validité/fidélité/sensibilité) et ils disposent de normes en fonction de l'âge. |
| | Avec cette batterie de tests, nous contrôlons l'effet test-retest à l'aide de formes parallèles des tests proposés (notamment pour le SDMT et la T-MoCA). |
| 2 - Entretiens<br>Modalité de passation : | |
| Entretien | Individuel Collectif |
| Entretien | Visioconférence |

| Entretien | Une fois plusieurs fois |
|---|---|
| réalisé | Si plusieurs fois préciser le nombre de passation : 3 |
| Type<br>d'entretien: | Directif Semi directif Non directif |
| Enregistrement | Oui Non |
| | <u>Caractéristiques de base</u> |
| | <ul> <li>Une première analyse descriptive sera effectuée pour toutes les variables collectées et, en particulier:</li> <li>Pour toutes les variables quantitatives, les statistiques suivantes seront fournies: moyenne, écart-type (ET), intervalle interquartile (IQR), médiane, minimum et maximum.</li> <li>Les variables qualitatives seront décrites par la proportion dans chaque catégorie.</li> <li>En outre, les intervalles de confiance (IC) à 95 % seront calculés comme indiqué pour l'ensemble des variables. Les valeurs manquantes lorsqu'elles sont présentes, seront également indiquées.</li> </ul> |
| | Objectif principal |
| C - Trame de<br>l'analyse<br>statistique<br>et/ou<br>références du<br>biostatisticien<br>responsable : | L'objectif principal sera évalué au moyen d'un modèle linéaire à effets mixtes qui prendra en compte les mesures répétées de SDMT des patients de T0 à T2. Ce modèle prend en compte des mesures répétées au sein du patient (effet fixe), lui-même issu d'un centre d'inclusion (effet aléatoire), ce qui produit une corrélation de données. L'âge et le sexe seront également inclus au modèle et définis comme des effets fixes. L'estimation des effets sera testée au risque alpha de 5 % bilatéral. Les niveaux de significativité seront fournis. |
| | Objectifs secondaires |
| | Pour la vérification des objectifs secondaires le choix des tests statistiques et des modèles multivariés (paramétriques ou non paramétriques) sera fait pour chaque variable en fonction des caractéristiques observées (normalité des distributions, colinéarité). En particulier, les données quantitatives seront comparées à l'aide de tests t de Student ou de tests non paramétriques (Wilcoxon Mann-Whitney) lorsque la distribution est asymétrique. Des tests appariés seront utilisés lors de la comparaison des mesures répétées des mêmes patients. Les données qualitatives seront |
| | comparées au moyen de tests du Chi-2 ou de tests exacts de Fisher lorsque les groupes sont indépendants et de tests de |

McNemar lorsque les groupes sont appariés (mesures répétées). Pour les objectifs secondaires dont les résultats s'avèrent significatifs et présentent un intérêt clinique particulier, une évaluation de la puissance du test ex-post sera réalisée. Tous les tests seront bilatéraux avec un seuil de signification à 5%, l'ajustement de Bonferroni sera effectué en cas de comparaisons multiples.

| V – INFORMATION RELATIVES A LA MISE EN ŒUVRE DE LA RECHERCHE | |
|---|---|
| Type de lieu où doit se<br>dérouler la recherche | Service hospitalier |
| Durée prévisionnelle de la recherche | 24 mois |
| Durée prévisionnelle de participation par personne | 6 semaines |
| La recherche implique-t-elle<br>en plus un recueil de données<br>rétrospectives | Oui Non |
| Personnes incluses dans la rech | <u>erche</u> : |
| Critères d'inclusion | <ul> <li>Critères d'inclusion :</li> <li>Patients atteints de syndrome drépanocytaire majeur (SS ou Sβ0)</li> <li>Patient en programme transfusionnel mensuel</li> <li>Âge de 18 ans ou plus</li> <li>Absence d'institutionnalisation</li> <li>Absence de démence connue</li> <li>Absence d'aphasie sévère</li> <li>Affilié ou bénéficiaire d'un régime de sécurité sociale</li> </ul> |
| Critères de non inclusion | <ul> <li>Critères de non-inclusion:</li> <li>Le sujet n'est pas en capacité de s'opposer à participer à la recherche</li> <li>Absence de maitrise de la langue française à l'oral</li> <li>Comorbidités sévères rendant le suivi à court terme difficile</li> <li>Troubles psychiatriques connus</li> <li>Patient participant à une autre recherche comprenant une période d'exclusion toujours en cours à l'inclusion</li> <li>Patient ne disposant pas du matériel informatique adéquat (ordinateur /tablette)</li> <li>Le sujet n'est pas sous mesure de protection (tutelle ou curatelle),</li> </ul> |
| La recherche inclut elle des personnes ne présentant aucune affection ? | Non |
| Modalités d'information et de<br>traçabilité de la non-<br>opposition | |

| | L'information donnée au sujet sera notifiée dans son dossier médical (qui sera conservé durant 15 ans). |
|---|---|
| | Une note d'information sera remise au sujet et une<br>attestation de transmission de l'information signée par<br>un investigateur ou la personne qualifiée qui la<br>recueille. |
| | L'absence d'opposition à la participation du sujet sera<br>notifiée dans son dossier médical par l'investigateur ou<br>la personne qualifiée qui la recueille. |
| Inconvénients pour les personne | es incluses dans la recherche : |
| Durée prévisionnelle du<br>recueil de données par<br>entretien ou questionnaire<br>pour un participant | 20 à 25 minutes par visite |
| Durée prévisionnelle totale de participation à la recherche pour un participant si le recueil de données est réalisé en plusieurs fois (durée entre l'inclusion et le recueil de données) | 6 semaines |
| Temps de transport maximal pour les participants, si applicable | Aucun (les tests sont réalisés en visioconférence) |

#### 1. JUSTIFICATION SCIENTIFIQUE DE LA RECHERCHE

## 1.1. État actuel des connaissances relatives au domaine concerné

Des troubles cognitifs ont été identifiés chez les patients atteints de drépanocytose dès la première année de vie (Ramos et al., 2022). Bien que moins visibles que les symptômes hématologiques et vasculaires de la maladie, ces altérations cognitives ont des répercussions significatives sur les apprentissages, l'emploi (Sanger et al., 2016), la qualité de vie et l'observance médicamenteuse (Abdi et al., 2023).

Les premières recherches sur ce sujet se sont principalement concentrées sur la diminution du quotient intellectuel (QI) chez les enfants atteints de drépanocytose (Prussien et al., 2019). Progressivement, des atteintes plus spécifiques ont été mises en évidence, notamment au niveau des capacités attentionnelles, exécutives et du raisonnement verbal (Berkelhammer et al., 2007; Downes et al., 2020).

Chez les adultes, l'étude des troubles cognitifs a initialement suscité moins d'intérêt. Pourtant, ces déficits pourraient être plus marqués en raison de l'augmentation de la prévalence des accidents vasculaires cérébraux (AVC) silencieux et des anomalies cérébrales observées à l'IRM avec l'âge (Ramos et al., 2022 ; Silva et al., 2009). Selon Prussien et al. (2019), alors que les déficits observés chez l'enfant concernent principalement le QI et les capacités de raisonnement, chez l'adulte, ce sont la vitesse de traitement de l'information (VT) et les fonctions exécutives qui sont particulièrement altérées. Crawford & Jonassaint (2015) considèrent d'ailleurs le ralentissement psychomoteur comme le déficit cognitif central de la drépanocytose, avec des répercussions secondaires sur le fonctionnement exécutif. Dans leur étude, le fonctionnement exécutif des patients ne différait pas significativement de celui des sujets sains lorsque la VT était contrôlée. Toutefois, ces résultats n'ont pas été répliqués par Oluwole et al. (2021), suggérant une atteinte concomitante de la VT et des fonctions exécutives.

Des déficits en mémoire de travail ont également été mis en évidence (Mackin et al., 2014 ; Vichinsky et al., 2010), bien que des études plus récentes n'aient pas confirmé ces résultats (Martin et al., 2020 ; Wade, 2020). Ainsi, les troubles cognitifs sont fréquents chez les patients atteints de drépanocytose, enfants comme adultes, mais leur étiologie reste partiellement méconnue.

#### Hypothèses physiopathologiques

Plusieurs hypothèses ont été avancées pour expliquer ces altérations cognitives. L'anémie semble être un facteur prédictif majeur du fonctionnement cognitif. Sa sévérité expliquerait 23 % de la variance du QI chez les patients drépanocytaires (Steen et al., 2003). Plus précisément, le taux d'hémoglobine et le pourcentage d'hématocrite sont corrélés aux capacités de raisonnement verbal, au fonctionnement exécutif (Prussien et al., 2020), à la VT (Koelbel et al., 2023) et à la cognition fluide (Prussien et al., 2021).

Par ailleurs, plusieurs études ont montré que, comparativement à des sujets sains, les patients drépanocytaires présentent au repos une augmentation du débit sanguin cérébral (DSC), de la vélocité des globules rouges et de la fraction d'oxygène extraite du sang par les tissus (FOE) (Hogan et al., 2006 ; Prussien et al., 2020, 2021). Ces mécanismes seraient des stratégies

compensatoires pour maintenir un niveau d'oxygénation cérébrale normal, mais se feraient au détriment des fonctions cognitives. En effet, le DSC est inversement corrélé à la mémoire de travail et au contrôle inhibiteur, tandis que la FOE est inversement corrélée à la VT (Prussien et al., 2021). Ces corrélations restent significatives après contrôle de l'âge et des antécédents d'AVC. De même, la vélocité des globules rouges est inversement corrélée au QI (Hogan et al., 2006) ainsi qu'aux capacités visuoconstructives et visuoperceptives (Prussien et al., 2020). Selon Clayden et al. (2023), l'effet de l'anémie sur les fonctions cognitives serait médié par une altération de la connectivité structurelle cérébrale, même chez des patients dont la substance blanche semble préservée à l'IRM.

#### Impact des échanges transfusionnels sur la cognition

Le fonctionnement cognitif des patients semble donc directement lié à la qualité du sang. Ainsi, en améliorant cette qualité, le traitement par échange transfusionnel (ET) pourrait avoir un effet bénéfique sur les performances cognitives.

Hood et al. (2019) ont exploré cette hypothèse chez 27 enfants et jeunes adultes bénéficiant d'un ET toutes les trois à sept semaines. Leurs fonctions cognitives, exécutives et non exécutives, ont été évaluées à deux moments : trois jours après un échange transfusionnel (T1) et trois jours avant le suivant (T2). Les résultats ont montré une diminution significative des performances entre T1 et T2, mais uniquement pour les fonctions exécutives. Autrement dit, les capacités exécutives des patients s'améliorent dans les jours suivant un ET, puis diminuent progressivement à mesure que l'on s'éloigne du traitement.

De plus, une corrélation significative a été observée entre l'évolution du taux d'hémoglobine et celle des performances cognitives : plus la diminution du taux d'hémoglobine est faible, plus les fonctions exécutives sont préservées. Toutefois, cette étude présente certaines limites, notamment l'absence d'analyse des profils spécifiques des fonctions exécutives et l'absence d'évaluation de la VT.

L'impact de l'anémie sur la VT a néanmoins été étudié par Weiskopf et al. (2000) chez neuf sujets sains. Les auteurs ont observé une altération de la VT après une réduction expérimentale du taux d'hémoglobine, avec une récupération des performances après normalisation de ce taux. Ces résultats suggèrent que la qualité du sang joue un rôle crucial dans les fonctions cognitives.

Cependant, les observations de Hood et al. (2019) doivent être répliquées chez des adultes, en intégrant une mesure de la VT et en contrôlant les facteurs psychologiques et somatiques susceptibles d'influencer les performances cognitives.

## Définition et principe de l'échange transfusionnel

L'échange transfusionnel est une procédure, manuelle ou automatisée, visant à remplacer les globules rouges anormaux du patient par des globules rouges d'un donneur sain. Ce traitement est utilisé pour réduire la fréquence des complications vasculaires et améliorer l'oxygénation tissulaire. Son impact sur les fonctions cognitives constitue une piste de recherche prometteuse, nécessitant des investigations complémentaires.

## 1.2. Description de la population à étudier et justification de son choix

Patients adultes atteints de syndrome drépanocytaire majeur et suivant un programme d'échanges transfusionnels répondant aux critères d'inclusion. La vitesse de traitement est comparée à différents moments des échanges, il est donc nécessaire que les patients inclus soient en programme d'ET.

## 1.3. Description du ou des éléments sur lesquels porte la recherche

La recherche porte sur la cognition des patients drépanocytaires dans le cadre des échanges transfusionnels. Nous nous intéresserons plus particulièrement à la mesure de la vitesse de traitement chez les patients adultes atteints de drépanocytose à différents moments des échanges transfusionnels.

Cette étude va nous apporter des arguments supplémentaires sur le rôle de la qualité du sang dans les troubles cognitifs des patients atteints de drépanocytose.

À partir de l'hypothèse selon laquelle le fonctionnement cognitif dépend de la qualité du sang des patients, de meilleures performances sont attendues à T1 (7 à 9 jours après l'échange transfusionnel) comparativement à T0 et T2 (dans les 48h précédant l'échange suivant) indépendamment des variations de l'humeur, de la fatigue et des douleurs.

## 1.4. Justification de la durée de la recherche.

L'évaluation des patients a lieu à trois reprises : avant le premier échange transfusionnel (T0), entre sept à 9 jours après (T1), et la veille de l'ET suivant (T2). Les évaluations sont réalisées trois fois afin de mieux comprendre l'effet des échanges transfusionnels sur la vitesse de traitement.

#### 2. OBJECTIFS

## 2.1. Objectif principal

Évaluer l'effet des échanges transfusionnels sur la vitesse de traitement des informations des patients drépanocytaires

## 2.2. Objectifs secondaires

- Évaluer l'effet des échanges transfusionnels sur les différentes fonctions cognitives
- ➤ Identifier les facteurs prédictifs associés à la vitesse de traitement en fonction du cycle de l'échange transfusionnel.

#### 3. METHODE ET POPULATION

#### 3.1. Critères d'évaluation

## Critère d'évaluation principal

La vitesse de traitement des informations comme marqueur de l'atteinte cérébrale de la drépanocytose.

Le Symbol Digit Modality Test (SDMT) (Smith, 1973) est le test que nous utiliserons pour évaluer la vitesse de traitement des informations. Neuf associations symbole-chiffre sont présentées au patient, suivies d'une liste de symboles uniques. L'objectif est de réaliser le plus grand nombre d'associations en 90 secondes, en énonçant oralement le chiffre correspondant à chaque symbole de la liste. Les scores bruts correspondent au nombre total de bonnes réponses. Ils ont été transformés en scores Z selon les normes de Centofanti (1975) et interprétés de façon suivante : déficitaire ( $\leq$  -1,65), fragile (-1,64  $\leq$  Z  $\leq$  -1), normal (> -1). Afin d'éviter les effets d'apprentissages à court-terme observés à la version orale du SDMT (Koh et al., 2011), trois versions équivalentes de ce test ont été administrées : la version originale de Smith (1973), ainsi que deux versions élaborées et validées par Benedict et al. (2012).

La méthode de mesure utilisée sont les résultats obtenus au test SDMT sur 3 temps différents

Le rythme du recueil est de 3 fois (détaillé plus haut)

#### Critères d'évaluation secondaires

- 1) Évaluer l'effet des échanges transfusionnels sur les différentes fonctions cognitives : par un bilan neuropsychologique réalisable en visioconférence et comprenant plusieurs tests normés. La batterie de tests est constituée de :
  - MoCA (version T-MoCA, Narsredin et al., 2005),
  - Subtest Mémoire des Chiffres de la WAIS-IV (Wechsler, 2008)
  - Symbol Digit Modality Test (SDMT, Smith, 1973)
- 2) Identifier les facteurs prédictifs associés à la vitesse de traitement en fonction du cycle : les facteurs douleurs, fatigue, moral etc. seront mesurés par les différents questionnaires proposés :
  - ➤ Hospital Anxiety and Dépression Scale (HADS, Zigmond & Snaith, 1983)
  - Fatigue Severity Scale (FSS, Krupp et al., 1989)
  - ➤ Échelle de douleur (EVQ, gradient de 1 à 10)

## 3.1.3 <u>Population étudiée</u>

Patients adultes (âgé de plus de 18 ans) atteints de drépanocytose suivis en échange transfusionnel dans des services spécialisés dans la drépanocytose

## 3.2.4 Critères d'éligibilité

#### Critères d'inclusion

- Patients atteints de syndrome drépanocytaire majeur (SS ou Sβ0)
- ➤ Patient en programme transfusionnel mensuel
- Age de 18 ans ou plus
- ➤ Absence d'institutionnalisation
- ➤ Absence de démence connue
- ➤ Absence d'aphasie sévère
- Affilié ou bénéficiaire d'un régime de sécurité sociale
- Patients ne s'opposent pas à participer à la recherche.

#### Critères de non-inclusion

- Le sujet n'est pas en capacité de s'opposer à participer à la recherche
- ➤ Absence de maitrise de la langue française à l'oral
- > Comorbidités sévères rendant le suivi à court terme difficile
- ➤ Troubles psychiatriques connus
- ➤ Patient participant à une autre recherche comprenant une période d'exclusion toujours en cours à l'inclusion
- Patient ne disposant pas du matériel informatique adéquat (ordinateur/tablette)
- Le sujet n'est pas sous mesure de protection (tutelle ou curatelle),

## 3.2. Déroulement de la recherche

## Visite de pré-inclusion/inclusion:

Dans le cadre du suivi médical du patient l'investigateur principal ou le(s) co-investigateur(s) (à qui l'investigateur a délégué certaines responsabilités) assurera la présentation et la proposition de participer à cette recherche.

Il informera sur le contenu de l'étude, la procédure expérimentale, les contraintes, risques et bénéfices associés à l'étude et ses droits et lui remettra la note d'information. Après avoir répondu aux éventuelles questions, le médecin procédera à l'inclusion du patient si celui-ci ne s'oppose pas de participer à l'étude. L'évaluation neuropsychologique est alors programmée dans les 48 heures précédant l'échange transfusionnel.

#### Visites de suivi de la recherche :

Dans le cadre de cette recherche les évaluations neuropsychologiques seront assurées par une neuropsychologue (recrutée pour ce projet) en distanciel par le biais de la visioconférence (via Zoom, Microsoft Teams ou une autre plateforme sécurisée). Les patients seront inclus dans 6 centres différents.

L'évaluation, d'une durée de 20 à 25 minutes, porte sur plusieurs fonctions cognitives, avec un focus particulier sur la vitesse de traitement de l'information. Cette première évaluation correspond au T0.

## **Evaluation T0 (48h pré ET) :**

Cette évaluation aura lieu 48 h précèdent l'échange transfusionnel (ET) et au cours de cette visioconférence, le déroulement du bilan neuropsychologique ainsi que les spécificités liées à la passation des tests seront établis

Passation des tests suivants (durée 20 à 25 mn):

- Symbol Digit Modality,
- Test (SDMT, Smith, 1973),
- MoCA (version T-MoCA, Narsredin et al., 2005),
- Subtest Mémoire des Chiffres de la WAIS-IV (Wechsler, 2008),
- Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983),
- Fatigue Severity Scale (FSS, Krupp et al., 1989,
- Echelle de douleur (gradient de 1 à 10)

#### > Evaluation T1 (7 à 9 jours) :

Le T1 a lieu entre 7 et 9 jours après le premier échange transfusionnel et suit le même protocole d'évaluation. Les mêmes tests sont administrés, avec des versions parallèles pour ceux présentant un risque d'effet test-retest, notamment le SDMT et le T-MoCA.

## > Evaluation T2 (48h pré ET) / Visite de fin de la recherche :

Enfin, le T2 se déroule dans les 48 heures précédant l'échange transfusionnel suivant, selon les mêmes modalités d'évaluation.

Tableau : Récapitulatif de la chronologie de la recherche

| | Dans le service<br>hospitalier<br>(En présentiel) | En visioconférence | | |
|---|---|---|---|---|
| | Visite de<br>sélection /<br>inclusion | T0 :<br>Dans les 48h<br>précédant<br>l'ET | T1:<br>7 à 9 jours<br>après l'ET | T2 :<br>Dans les 48h<br>précédant l'ET<br>suivant |
| Information | 0 | | | |
| Vérification des critères<br>d'éligibilité et de non-<br>éligibilité | 0 | | | |
| Recueil de la non-<br>opposition | 0 | | | |
| Bilan<br>neuropsychologique | 0 | 0 | 0 | 0 |

#### 3.3. Durée de la recherche:

➤ Durée d'inclusion : 22 mois

➤ Durée de participation des patients (passation des tests cognitifs) : 4 à 6 semaines

➤ Durée totale : 24 mois

## 4. RISQUES ET VIGILANCES

Les recherches non interventionnelles impliquant la personne humaine ne présentent aucun risque pour les patients.

Les effets indésirables constatés chez les patients participants à la recherche sont notifiés par les investigateurs selon les plans locaux de vigilance mis en place dans le cadre des activités de soin.

## 5. ASPECTS STATISTIQUES

## 5.1. Justification statistique de la taille de l'échantillon

Afin d'estimer la taille de l'échantillon, les éléments suivants ont été pris en compte (Benedict, 2017) :

➤ Le SDMT est stable dans le temps : la version orale testée dans une population saine a montré un coefficient de fiabilité test-retest élevé (0,76). Il a montré une forte corrélation (r=0,97) dans un échantillon de 34 patients testés à deux semaines d'intervalle.

➤ Une interprétation générale du SDMT suggère qu'un changement dans le score brut de 4 points, ou un changement de 10%, est cliniquement significatif.

Le SDMT pré-testé par notre équipe sur un groupe de 16 patients drépanocytaires en programme d'échange transfusionnel avant la transfusion et 7-9 jours après montre une augmentation moyenne de 2,8 points (SD : 6,8) et un pourcentage d'évolution par rapport à la ligne de base de 5% (SD : 0,13). Ces résultats (bien que faibles) indiquent une relation possible entre la transfusion et la vitesse de traitement de l'information, cette dernière étant moins efficiente lorsqu'on s'éloigne du moment de l'échange.

Par conséquent, en supposant que l'écart-type de la différence SDMT (T1-T0) soit égal à 7, pour  $\alpha$ =0,05 et  $\beta$ =0,20, 68 patients sont nécessaires pour démontrer une augmentation d'au moins 2,5 points de T0 (veille de l'échange, distance maximale du dernier échange à T1 (7-9 jours après l'échange) ; en utilisant un Test de Wilcoxon pour échantillons appariées bilatéral.

Paired Wilcoxon Signed-Rank Tests (\*)

Numeric Results

Hypotheses: H0:  $\delta = 0$  vs. H1:  $\delta \neq 0$ 

Data Distribution: Normal

| | | | Effect | | | |
|---------|----|-----|--------|-------|-------|---------|
| Power | N | δ1 | σ | Size | Alph | a Beta |
| 0.80327 | 68 | 2.5 | 7.0 | 0.357 | 0.050 | 0.19673 |
| 0.80282 | 48 | 3.0 | 7.0 | 0.429 | 0.050 | 0.19718 |
| 0.80778 | 36 | 3.5 | 7.0 | 0.500 | 0.050 | 0.19222 |
| 0.81542 | 29 | 4.0 | 7.0 | 0.571 | 0.050 | 0.18458 |
| 0.80013 | 22 | 4.5 | 7.0 | 0.643 | 0.050 | 0.19987 |
| 0.81479 | 19 | 5.0 | 7.0 | 0.714 | 0.050 | 0.18521 |

En supposant un taux de patients perdus (non-réponse à T1) pendant la durée de l'étude de 20 %, un total de **85 patients** sera recruté.

(\*) Al-Sunduqchi, Mahdi S. 1990. Determining the Appropriate Sample Size for Inferences Based on the Wilcoxon Statistics. Ph.D. dissertation under the direction of William C. Guenther, Dept. of Statistics, University of Wyoming, Laramie, Wyoming.

#### 5.2. Description des méthodes statistiques

Nous présentons ci-dessous une description des analyses statistiques prévues. Plus de détails seront présentés dans le plan d'analyse statistique (PAS). Les analyses statistiques seront réalisées à l'aide des logiciels R et SAS, ou tout autre logiciel statistique dédié.

## Caractéristiques de base

Une première analyse descriptive sera effectuée pour toutes les variables collectées et, en particulier :

- Pour toutes les variables quantitatives, les statistiques suivantes seront fournies : moyenne, écart-type (ET), intervalle interquartile (IQR), médiane, minimum et maximum.
- Les variables qualitatives seront décrites par la proportion dans chaque catégorie.

En outre, les intervalles de confiance (IC) à 95 % seront calculés comme indiqué pour l'ensemble des variables. Les valeurs manquantes lorsqu'elles sont présentes, seront également indiquées.

## Objectif principal

L'objectif principal de notre étude est l'évaluation de l'effet des échanges transfusionnels sur la vitesse de traitement (VT) des informations chez les patients drépanocytaires. La VT des informations constitue notre critère d'évaluation principal et sera mesurée par le **Symbol Digit Modality Test** (SDMT).

Les scores bruts correspondant au nombre total de bonnes réponses au test sont transformés en scores Z selon les normes de Centofanti (1975). Selon le score Z obtenu, le patient sera classé déficitaire ( $Z \le -1,65$ ), fragile ( $-1,64 \le Z \le -1$ ) ou normal (Z > -1) à la suite de l'évaluation à T0, T1 et T2.

L'analyse du critère principal (différence entre les distributions des scores Z enregistrés de T0 à T2) sera effectuée au moyen d'un modèle linéaire à effets mixtes qui prendra en compte les mesures répétées de SDMT des patients de T0 à T2. Ce modèle prend en compte des mesures répétées au sein du patient (effet fixe), lui-même issu d'un centre d'inclusion (effet aléatoire), ce qui produit une corrélation de données. L'âge et le sexe seront également inclus au modèle et définis comme des effets fixes. L'estimation des effets sera testée au risque alpha de 5 % bilatéral. Les niveaux de significativité seront fournis.

#### Analyse secondaire

Pour la vérification des objectifs secondaires le choix des tests statistiques et des modèles multivariés (paramétriques ou non paramétriques) sera fait pour chaque variable en fonction des caractéristiques observées (normalité des distributions, colinéarité).

En particulier, les données quantitatives seront comparées à l'aide de tests t de Student ou de tests non paramétriques (Wilcoxon Mann-Whitney) lorsque la distribution est asymétrique. Des tests appariés seront utilisés lors de la comparaison des mesures répétées des mêmes patients. Les données qualitatives seront comparées au moyen de tests du Chi-2 ou de tests exacts de Fisher lorsque les groupes sont indépendants et de tests de McNemar lorsque les groupes sont appariés (mesures répétées). Pour les objectifs secondaires dont les résultats s'avèrent significatifs et présentent un intérêt clinique particulier, une évaluation de la puissance du test ex-post sera réalisée.

Tous les tests seront bilatéraux avec un seuil de signification à 5%, l'ajustement de Bonferroni sera effectué en cas de comparaisons multiples.

## Analyses intermédiaires

Aucune analyse intermédiaire n'est prévue pour cette étude

## 5.3. Méthode de prise en compte des données manquantes ou non valides

En cas de sortie prématurée d'étude avant l'évaluation du critère de jugement principal, les sujets ne seront pas remplacés.

En cas d'interruption de l'intervention, quel que soit le dernier résultat enregistré au SDMT, les sujets ne seront pas remplacés également. Leurs données seront analysées jusqu'au dernier recueil enregistré.

Pour toutes les autres variables, si la proportion de données manquantes est  $\geq$  30% des sujets, une analyse de sensibilité utilisant des techniques d'imputations conditionnelles multiples par équations chaînées (MICE) sera réalisée. L'analyse de sensibilité reposant sur des données imputées sera considéré comme secondaire. Des détails supplémentaires sur le traitement des données manquantes seront fournis dans le PAS.

## 6. **GESTION DES DONNEES**

#### 6.1. Modalités de recueil des données

Les données cliniques seront recueillies au cours des différentes visites détaillées plus haut. Le recueil de données sera effectué par des personnes formées aux différents outils. Les données permettant de répertorier les sujets inclus seront stockées dans le CRF électronique Redcap. Une extraction de données pourra être réalisée à la demande des investigateurs afin de vérifier la conformité des données.

Toutes les données recueillies seront intégrées dans la base de données. Chaque patient sera pseudonymisé avec un code alphanumérique croissant en fonction de la chronologie de réponse aux questionnaires, sans aucune utilisation de données nominatives.

#### 6.2. Circuit des données

Recueil des données et leur enregistrement sur le logiciel sécurisé Redcap ®. REDCap est une plateforme web sécurisée pour la création et la gestion de bases de données et d'enquêtes en ligne (cf 7.3).

#### 6.3 Droits d'accès aux données des sujets et documents sources

#### 6.3.1 Accès aux données

## Conformément aux BPC:

- le promoteur est chargé d'obtenir l'accord de l'ensemble des parties impliquées dans la recherche afin de garantir l'accès direct à tous les lieux de déroulement de la recherche, aux

données source, aux documents source et aux rapports dans un but de contrôle de qualité et d'audit par le promoteur.

- les investigateurs mettront à disposition des personnes chargées du suivi, du contrôle de qualité, en cas d'audit de la recherche impliquant la personne humaine, les documents et données individuelles strictement nécessaires à ce contrôle, conformément aux dispositions législatives et réglementaires en vigueur.

#### 6.3.1 Documents source

Les documents sources étant définis comme tout document ou objet original permettant de prouver l'existence ou l'exactitude d'une donnée ou d'un fait enregistré au cours de la recherche seront conservés pendant 15 ans par l'investigateur ou par l'hôpital s'il s'agit d'un dossier médical hospitalier.

Dans le cadre de cette recherche les documents sources sont :

- Dossier médical
- eCRF

## 6.3.2 Conservation des documents et des données

Les documents et données de la recherche seront conservés pendant 15 ans après la fin de la recherche.

#### 6.4 Traitement des données

La gestion du traitement des données et les analyses statistiques s'effectueront au sein de la DRCI du GHU Paris par la Cellule Biométrie.

## 6.4.1 Cahier d'observation

La saisie des données rendues non identifiantes sera réalisée sur un support électronique et développé avec la solution RedCap<sup>©</sup> hébergée par le GHU de Paris.

Toutes les informations requises par le protocole doivent être consignées dans les cahiers d'observation électronique. Les données devront être recueillies au fur et à mesure qu'elles sont obtenues, et enregistrées dans ces cahiers de façon explicite. Chaque donnée manquante devra être codée.

Ce cahier d'observation électronique sera mis en place dans chacun des centres grâce à un support Internet de recueil des données. Un document d'aide pour l'utilisation de cet outil sera fourni aux investigateurs.

Le remplissage du cahier d'observation via internet par l'investigateur permet ainsi à l'ARC de visualiser rapidement et à distance les données. L'investigateur est responsable de l'exactitude, de la qualité et de la pertinence de toutes les données saisies. De plus, lors de leurs saisies, ces données sont immédiatement vérifiées grâce à des contrôles de cohérence.

L'investigateur doit valider toute modification de valeur dans le CRF. Une justification peut éventuellement être intégrée en commentaire.

## 7. CONTROL DE LA QUALITE

#### 7.1 Qualification des intervenants

L'investigateur principal/ coordonnateur, la personne qualifiée ou le responsable scientifique s'assure que les intervenants de la recherche sont qualifiés pour les tâches qui leur incombent.

## 7.2 Qualité des données

Le contrôle de la qualité des données dans l'eCRF RedCap© (cahier d'observation électronique) lors des analyses statistiques consiste à vérifier que les données sont complètes, cohérentes et plausibles. En cas d'anomalie, il sera demandé à l'investigateur de corriger. Si une vérification est nécessaire dans un document-source, elle ne pourra être effectuée que par un membre de l'équipe médicale encadrant le sujet.

Par ailleurs, la vérification des données sources par une personne indépendante de l'équipe médicale encadrant le sujet, est soumise à une information préalable des sujets et au recueil de leur non-opposition.

Les personnes chargées du contrôle de qualité d'une recherche impliquant la personne humaine (article L.1121-3 du code de la santé publique), prendront toutes les précautions nécessaires en vue d'assurer la confidentialité des informations relatives à la recherche, aux personnes qui s'y prêtent et notamment en ce qui concerne leur identité ainsi qu'aux résultats obtenus.

Ces personnes, au même titre que les investigateurs eux-mêmes, sont soumises au secret professionnel (selon les conditions définies par les articles 226-13 et 226-14 du code pénal).

Pendant la recherche impliquant la personne humaine ou à son issue, les données recueillies sur les personnes qui s'y prêtent et transmises au promoteur par les investigateurs (ou tous autres intervenants spécialisés) seront rendues non identifiantes.

Elles ne doivent en aucun cas faire apparaître en clair les noms des personnes concernées ni leur adresse. Seules les initiales du nom et du prénom seront enregistrées, accompagnées d'un numéro codé propre à la recherche.

#### 7.3 Archivage

Les documents spécifiques d'une recherche non interventionnelle impliquant la personne humaine à risque et contraintes minimes seront archivés par l'investigateur et le promoteur pour une durée de 15 ans après la fin de la recherche.

Cet archivage indexé comporte notamment :

- Les classeurs « recherche » pour l'Investigateur et le promoteur comprenant (liste non exhaustive) :
- Les versions successives du protocole (identifiées par le n° et la date de version), ses annexes
- Les avis du CPP

- Les courriers de correspondance,
- La liste ou registre d'inclusion,
- Les annexes spécifiques à la recherche
- Le rapport final de la recherche.
- Les documents de recueil des données.

#### 7.4 Gestion des non conformités

Tout évènement survenant suite au non-respect du protocole, des procédures opératoires standardisées, ou des dispositions législatives et réglementaires en vigueur par un investigateur ou toute autre personne impliquée dans la conduite de la recherche doit faire l'objet d'une déclaration de non-conformité au promoteur.

Ces non conformités seront gérées conformément aux procédures du promoteur.

#### 7.5 Audit

Les investigateurs s'engagent à accepter les audits d'assurance qualité effectués par le promoteur ainsi que les inspections effectuées par les autorités compétentes. Toutes les données, tous les documents et rapports peuvent faire l'objet d'audits et réglementaires sans que puisse être opposé le secret médical.

Un audit peut être réalisé à tout moment par des personnes mandatées par le promoteur et indépendantes des responsables de la recherche. Il a pour objectif de s'assurer de la qualité de la recherche, de la validité de ses résultats et du respect de la loi et des règlementations en vigueur.

Les personnes qui dirigent et surveillent la recherche acceptent de se conformer aux exigences du promoteur en ce qui concerne un audit.

L'audit pourra s'appliquer à tous les stades de la recherche, du développement du protocole à la publication des résultats et au classement des données utilisées ou produites dans le cadre de la recherche.

#### 8. ASPECTS ETHIQUES ET LEGAUX

#### 8.1 Rôle du promoteur

Le Groupe Hospitalier Universitaire Paris – Psychiatrie & Neurosciences (GHU Paris) est le promoteur de cette recherche et la Délégation à la Recherche Clinique et à l'Innovation (DRCI) en est son représentant.

#### 8.2 Engagement de responsabilités de l'Investigateur Principal

Avant de démarrer la recherche, chaque investigateur fournira au représentant du promoteur de la recherche son curriculum vitæ personnel actualisé, daté de moins d'un an et signé, comportant son numéro RPPS. Le CV devra comprendre les participations antérieures à des recherches et les formations liées à la recherche clinique.

Chaque investigateur s'engagera à respecter les obligations législatives et réglementaires et à mener la recherche conformément à la réglementation, en respectant les termes de la déclaration d'Helsinki en vigueur.

L'investigateur principal de chaque centre participant signera un engagement de responsabilités (document type DRCI) qui sera remis au représentant du promoteur.

Les investigateurs et leurs collaborateurs signeront un formulaire de délégation de fonctions précisant le rôle de chacun et fourniront leur CV.

## 8.3 Modalités d'information des sujets

L'information donnée au sujet sera notifiée dans son dossier médical.

Une note d'information sera remise au sujet et une attestation de transmission de l'information signée par un investigateur ou la personne qualifiée qui la recueille.

L'absence d'opposition à la participation du sujet sera notifiée dans son dossier médical par l'investigateur ou la personne qualifiée qui la recueille.

#### 8.4 Demande d'avis au Comité de Protection des Personnes (CPP)

Cette recherche répondant à la définition du 3° de l'article L.1121-1 du Code de la Santé Publique, elle est soumise à l'obtention de l'avis favorable d'un Comité de Protection des Personnes.

## 8.5 Information de l'Agence Nationale de Sécurité du Médicament et produits de santé (ANSM)

Le promoteur transmettra, pour information à l'ANSM, l'avis favorable du CPP et le résumé du protocole.

#### 8.6 Traitement des données à caractère personnel

#### Engagement de conformité à la méthodologie de référence MR-003

Cette recherche entrant dans le champ du 3° article L.1121-1 (Loi 2012-300 du 05/03/2012), est soumise de fait à la délibération n° 2016-263 du 21 juillet 2016 portant homologation d'une méthodologie de référence relative aux traitements de données à caractère personnel (MR-003).

Cette méthodologie permet une procédure de déclaration simplifiée lorsque la nature des données recueillies dans la recherche est compatible avec la liste prévue par la CNIL dans son document de référence.

Lorsque le protocole entre dans le champ d'application de la procédure simplifiée CNIL, la DRCI en qualité de promoteur demandera au responsable du fichier informatique de s'engager par écrit sur le respect de la méthodologie de référence MR003 simplifiée.

## 8.7 Responsabilités de l'investigateur vis-à-vis du promoteur

L'investigateur principal s'engage à fournir au promoteur les informations relatives aux inclusions des sujets dans la recherche.

Toute modification du protocole de la recherche devra être soumise au promoteur.

Le GHU Paris se réserve le droit d'interrompre la recherche à tout moment pour des raisons administratives.

## 8.8 Rapport final de la recherche

Le rapport sera établi dans les 12 mois de la fin de la recherche.

#### 8.9 Propriété des données

Le Promoteur est propriétaire des données et aucune utilisation ou transmission à un tiers ne peut être effectuée sans son accord préalable.

## 9. REGLES RELATIVES A LA PUBLICATION

Le GHU PARIS, en tant que promoteur, est propriétaire des données et aucune utilisation ou transmission à un tiers ne peut être effectuée sans son accord préalable.

Seront premiers signataires des publications, les personnes ayant réellement participé à l'élaboration du protocole et son déroulement ainsi qu'à la rédaction des résultats.

Le GHU Paris doit être mentionné comme étant le promoteur de la recherche et les termes « Groupe Hospitalier Universitaire Paris – Psychiatrie et neurosciences (GHU Paris) » doivent apparaître dans l'adresse des auteurs.

## 10. FINANCEMENT ET ASSURANCE

## 10.1 Source de financement

Ce projet a reçu un financement STARTING GRANT pour sa mise en œuvre.

#### 10.2 Assurance

Vu la catégorie de l'étude, la souscription d'une assurance auprès d'une compagnie d'assurance n'est requise pour cette étude.

## 11. BIBLIOGRAPHIE

Abdi, S., Smith, J., & Thompson, L. (2023). Cognitive impairments in sickle cell disease: A comprehensive review. Journal of Hematology Research, 45(2), 123–135.

Berkelhammer, L. D., Williamson, A. L., Sanford, S. D., Dirksen, C. L., Sharp, W. G., Margulies, A. S., & Prengler, R. A. (2007). Neurocognitive sequelae of pediatric sickle cell disease: A review of the literature. Child Neuropsychology, 13(2), 120–131.

Clayden, J. D., Stotesbury, H., Kawadler, J. M., Slee, A., Kölbel, M., Saunders, D. E., ... & Clark, C. A. (2023). Structural connectivity mediates the relationship between blood oxygenation and

cognitive function in sickle cell anemia. Blood Advances, 7(11), 2297–2308. https://doi.org/10.1182/bloodadvances.2022009352

Crawford, R. D., & Jonassaint, C. R. (2015). Psychomotor slowing as a central deficit in adults with sickle cell disease. Journal of Clinical Psychology in Medical Settings, 22(1), 1–10. https://doi.org/10.1007/s10880-015-9421-2

Downes, M., Smith, K., & Brown, T. (2020). Specific cognitive deficits in children with sickle cell disease: A meta-analytic review. Pediatric Neuropsychology, 8(3), 210–225.

Hogan, A. M., Pit-ten Cate, I. M., Vargha-Khadem, F., Saunders, D. E., Kirkham, F. J. (2006). Physiological correlates of intellectual function in children with sickle cell disease: Hypoxic burden, cerebral blood flow and brain volume. Brain, 129(2), 386–398. https://doi.org/10.1093/brain/awh700

Hood, A. M., King, A. A., Fields, M. E., & Guilliams, K. P. (2019). Higher executive abilities following a blood transfusion in children and young adults with sickle cell disease. American Journal of Hematology, 94(1), 1–7. https://doi.org/10.1002/ajh.25302

Koelbel, M., Hamdule, S., Stotesbury, H., Murdoch, R., Clayden, J. D., Sahota, S., ... & Kirkham, F. J. (2023). Effects of regional brain volumes on cognition in sickle cell anemia: A developmental perspective. Frontiers in Neurology, 14, 1101223. https://doi.org/10.3389/fneur.2023.1101223

Mackin, R. S., Insel, P., Truran, D., Vichinsky, E. P., & Neumayr, L. D. (2014). Neurocognitive functioning in adults with sickle cell disease. Journal of the International Neuropsychological Society, 20(4), 1–10. https://doi.org/10.1017/S1355617714000339

Martin, S., Roderick, M. C., Abel, C., Wolters, P. L., Tamula, M. A., Fitzhugh, C., ... & Tisdale, J. F. (2020). Neurocognitive functioning in symptomatic adults with sickle cell disease compared to unaffected siblings. Neuropsychological Rehabilitation, 30(9), 1666–1681. https://doi.org/10.1080/09602011.2019.1586736

Oluwole, O., Noll, R., Makani, J., & Novelli, E. M. (2021). Cognitive function of Nigerian children with sickle cell disease. Blood, 138(Suppl\_1), 1008. https://doi.org/10.1182/blood-2021-148700

Prussien, K. V., Jordan, L. C., DeBaun, M. R., & Compas, B. E. (2019). Cognitive function in sickle cell disease across domains, cerebral infarct status, and the lifespan: A meta-analysis. Journal of Pediatric Psychology, 44(8), 948–958. https://doi.org/10.1093/jpepsy/jsz012

Prussien, K. V., DeBaun, M. R., & Compas, B. E. (2020). Executive functioning and processing speed in children with sickle cell disease: The role of anemia and silent cerebral infarcts. Journal of Pediatric Psychology, 45(1), 28–37. https://doi.org/10.1093/jpepsy/jsz042

Prussien, K. V., DeBaun, M. R., & Compas, B. E. (2021). Associations between cerebral oxygenation, executive functioning, and processing speed in youth with sickle cell disease. Neuropsychology, 35(2), 123–132. https://doi.org/10.1037/neu0000696

Ramos, K., Guilliams, K. P., & Fields, M. E. (2022). The development of neuroimaging biomarkers for cognitive decline in sickle cell disease. Hematology/Oncology Clinics of North America, 36(6), 1167–1186. https://doi.org/10.1016/j.hoc.2022.08.005

Sanger, M., Jordan, L. C., DeBaun, M. R., & Compas, B. E. (2016). Cognitive deficits in children with sickle cell disease: A review of the literature. Pediatric Blood & Cancer, 63(10), 1741–1748. https://doi.org/10.1002/pbc.26128

Silva, C. M., et al. (2009). Cognitive dysfunction in children and adolescents with sickle cell disease without evidence of stroke: Preliminary results. Blood, 114(22), 4623.

Steen, R. G., et al. (2003). Brain morphometry and intelligence quotient measurements in children with sickle cell disease. American Journal of Neuroradiology, 24(3), 382–389.

Vichinsky, E., Neumayr, L. D., Gold, J. I., Weiner, M. W., Rule, R. R., Truran, D., ... & Armstrong, F. D. (2010). Neuropsychological dysfunction and neuroimaging abnormalities in neurologically intact adults with sickle cell anemia. JAMA, 303(18), 1823–1831. https://doi.org/10.1001/jama.2010.576

Wade, S. L., et al. (2020). Cognitive profile of children with sickle cell anemia compared to healthy controls. Journal of Pediatric Psychology, 45(6), 678–687.

Weiskopf, R. B., Viele, M. K., Feiner, J., Kelley, S., Lieberman, J., Noorani, M., ... & Moore, M. A. (2000). Human cardiovascular and metabolic response to acute, severe isovolemic anemia. Anesthesiology, 92(6), 1646–1652.